CLINICAL TRIAL: NCT04979078
Title: Evaluating the Effectiveness of Photobiomodulation Therapy in the Management of Hand-foot Syndrome and Hand-foot Skin Reaction: A Single-arm Trial
Brief Title: Photobiomodulation Therapy in the Management of Hand-foot Syndrome and Hand-foot Skin Reaction
Acronym: DermLight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Collaborators: Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/071
Record Dates: First submitted 2021-07-16; First posted 2021-07-27 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Hand-foot Syndrome; Hand-foot Skin Reaction
Keywords: Dermatology; Oncology; Photobiomodulation; Skin toxicity; Hand-foot syndrome; Hand-foot skin reaction; Hand-foot skin toxicity; Supportive cancer care; Light therapy
MeSH Terms: conditions — Hand-Foot Syndrome; Neoplasms | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): The experimental group receives 9 sessions of photobiomodulation therapy (3x/week for 3 weeks).
  Interventions: Device: Photobiomodulation therapy (PBMT)

INTERVENTIONS:
Device: Photobiomodulation therapy (PBMT) — Patients will receive PBM on the sole of their feet and palms of their hands

SUMMARY:
Hand-foot syndrome (HFS) is a side effect of chemotherapy. HFS is characterized by redness, swelling, and pain on the palms of the hands and/or soles of the feet, which can progress to blistering. Hand-foot skin reaction (HFSR) refers to symptoms affecting the hands and/or feet associated with multikinase inhibitors (TKIs). HFS and HFSR are painful complications that can lead to compromised daily activities, sleep-wake disturbance and impaired mobility, eventually decreasing Quality of Life (QoL).

Photobiomodulation therapy (PBMT) is a non-invasive therapy based on the application of visible and/or near-infrared light produced by a laser diode or a light-emitting diode. The scientifically proven biologic effects of PBM are improved wound healing, and a reduction in pain, inflammation, and oedema. The aim of this study is to evaluate the effectiveness of PBMT in the management of HFS and HFSR.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the efficacy of PBMT in the management of HFS and HFSR in patients with cancer treated with chemotherapy or TKIs up to 2 weeks post-PBMT.

Primary objective: The study seeks primarily to determine the effectiveness of PBMT in reducing the severity of HFS and HFSR in patients with cancer of different etiology undergoing chemotherapy or TKIs, diagnosed with HFS or HFSR (grade 1-3).

Secondary objective 1 : HFS/HFSR-related symptoms

A secondary aim of this study is to evaluate if PBMT and can reduce the HFS/HSFR-related symptoms during PBM treatment and up to 2 weeks post-PBMT

Secondary Objective 2: Quality of life

A secondary aim of this study is to evaluate if PBMT can improve the patients' QoL during PBM treatment and up to 2 weeks post-PBMT

Secondary Objective 3: Patient satisfaction

A secondary aim of this study is to evaluate if patients are satisfied with PBMT as a treatment for HFS and HFSR during the treatment sessions and up to 2 weeks post-PBMT

Secondary Objective 4: PBM safety

A secondary aim of this study is to evaluate the safety of PBM in oncologic patients up to 5 years post-PBMT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer of different aetiologies
* Undergoing chemotherapy or targeted therapy (TKIs)
* Diagnosed with HFS-HFSR grade 1, 2 or 3 (National Cancer Institute - Common Terminology Criteria for Adverse Events, NCI-CTCAE v5)
* Age ≥ 18 years
* Able to comply to the study protocol
* Able to sign written informed consent

Exclusion Criteria:

* Pre-existing skin rash, ulceration or open wound in the treatment area (hand, foot)
* Known allergy to polyurethane
* Substance abuse patients or patients with medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results as judged by the investigator
* Any condition that is unstable or could affect the safety of the patient and their compliance in the study as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-12 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Skin reaction evaluation - CTCAE | Baseline
  The severity of the skin reactions will be evaluated by the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5.
Skin reaction evaluation - CTCAE | Session 3 of PBMT
  The severity of the skin reactions will be evaluated by the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5.
Skin reaction evaluation - CTCAE | Session 6 of PBMT
  The severity of the skin reactions will be evaluated by the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5.
Skin reaction evaluation - CTCAE | Final PBM session (session 9)
  The severity of the skin reactions will be evaluated by the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5.
Skin reaction evaluation - CTCAE | 2 weeks post-PBMT
  The severity of the skin reactions will be evaluated by the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5.
Skin reaction evaluation - WHO | Baseline
  The severity of the skin reactions will be evaluated by the World Health Association (WHO) grading scale for HFS/HFSR
Skin reaction evaluation - WHO | Session 3 of PBMT
  The severity of the skin reactions will be evaluated by the World Health Association (WHO) grading scale for HFS/HFSR
Skin reaction evaluation - WHO | Session 6 of PBMT
  The severity of the skin reactions will be evaluated by the World Health Association (WHO) grading scale for HFS/HFSR
Skin reaction evaluation - WHO | Final PBM session (session 9)
  The severity of the skin reactions will be evaluated by the World Health Association (WHO) grading scale for HFS/HFSR
Skin reaction evaluation - WHO | 2 weeks post-PBMT
  The severity of the skin reactions will be evaluated by the World Health Association (WHO) grading scale for HFS/HFSR
Clinical photograph | Baseline
  A clinical photograph of the palm of patients' hands and sole of their feet
Clinical photograph | Session 3 of PBMT
  A clinical photograph of the palm of patients' hands and sole of their feet
Clinical photograph | Session 6 of PBMT
  A clinical photograph of the palm of patients' hands and sole of their feet
Clinical photograph | Final PBM session (session 9)
  A clinical photograph of the palm of patients' hands and sole of their feet
Clinical photograph | 2 weeks post-PBMT
  A clinical photograph of the palm of patients' hands and sole of their feet

SECONDARY OUTCOMES:
Patient subjective evaluation of skin reactions | Baseline
  The patients will be asked to complete a questionnaire to evaluate the intensity of eight common symptoms of HFS/HFSR: pruritus, dryness, erythema, burning sensation, oedema, desquamation, blistering, and pain on an 11-point Numerical Rating Scale (NRS)
Patient subjective evaluation of skin reactions | Session 3 of PBMT
  The patients will be asked to complete a questionnaire to evaluate the intensity of eight common symptoms of HFS/HFSR: pruritus, dryness, erythema, burning sensation, oedema, desquamation, blistering, and pain on an 11-point Numerical Rating Scale (NRS)
Patient subjective evaluation of skin reactions | Session 6 of PBMT
  The patients will be asked to complete a questionnaire to evaluate the intensity of eight common symptoms of HFS/HFSR: pruritus, dryness, erythema, burning sensation, oedema, desquamation, blistering, and pain on an 11-point Numerical Rating Scale (NRS)
Patient subjective evaluation of skin reactions | Final PBM session (Session 9)
  The patients will be asked to complete a questionnaire to evaluate the intensity of eight common symptoms of HFS/HFSR: pruritus, dryness, erythema, burning sensation, oedema, desquamation, blistering, and pain on an 11-point Numerical Rating Scale (NRS)
Patient subjective evaluation of skin reactions | 2 weeks post-PBMT
  The patients will be asked to complete a questionnaire to evaluate the intensity of eight common symptoms of HFS/HFSR: pruritus, dryness, erythema, burning sensation, oedema, desquamation, blistering, and pain on an 11-point Numerical Rating Scale (NRS)
Quality of life - DLQI | Baseline
  Dermatology Life Quality Index (DLQI) is a questionnaire with 10 items and is used to measure QoL of dermatological patients.
Quality of life - DLQI | Session 3 of PBMT
  Dermatology Life Quality Index (DLQI) is a questionnaire with 10 items and is used to measure QoL of dermatological patients.
Quality of life - DLQI | Session 6 of PBMT
  Dermatology Life Quality Index (DLQI) is a questionnaire with 10 items and is used to measure QoL of dermatological patients.
Quality of life - DLQI | Final PBM session (session 9)
  Dermatology Life Quality Index (DLQI) is a questionnaire with 10 items and is used to measure QoL of dermatological patients.
Quality of life - DLQI | 2 weeks post-PBMT
  Dermatology Life Quality Index (DLQI) is a questionnaire with 10 items and is used to measure QoL of dermatological patients.
Quality of life - Skindex-29 | Baseline
  The skindex-29 is a validated instrument to measures patients' QoL specifically correlated with skin conditions. It has 3 scales addressing emotions (10 items), symptoms (7 items) and functioning (12 items).
Quality of life - Skindex-29 | Session 3 of PBMT
  The skindex-29 is a validated instrument to measures patients' QoL specifically correlated with skin conditions. It has 3 scales addressing emotions (10 items), symptoms (7 items) and functioning (12 items).
Quality of life - Skindex-29 | Session 6 of PBMT
  The skindex-29 is a validated instrument to measures patients' QoL specifically correlated with skin conditions. It has 3 scales addressing emotions (10 items), symptoms (7 items) and functioning (12 items).
Quality of life - Skindex-29 | Final PBM session (session 9)
  The skindex-29 is a validated instrument to measures patients' QoL specifically correlated with skin conditions. It has 3 scales addressing emotions (10 items), symptoms (7 items) and functioning (12 items).
Quality of life - Skindex-29 | 2 weeks post-PBMT
  The skindex-29 is a validated instrument to measures patients' QoL specifically correlated with skin conditions. It has 3 scales addressing emotions (10 items), symptoms (7 items) and functioning (12 items).
Patients' satisfaction with the therapeutic intervention | Final PBM session (session 9)
  The patients will be asked to evaluate their satisfaction with PBM on a 5-point Likert scale
Patients' satisfaction with the therapeutic intervention | Two weeks post-PBMT
  The patients will be asked to evaluate their satisfaction with PBM on a 5-point Likert scale

OTHER OUTCOMES:
General patient-, disease-, and treatment-related information | Baseline
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (i.e., gender, age, smoking history, work habits, physical activity, skin condition, alcohol use, and medication use). Furthermore, information about disease- and treatment-related risk factors will be collected through medical records (e.g., tumor type and stage, tumor site, treatment type, etc).
General patient-, disease-, and treatment-related information | Final PBM session (session 9)
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (i.e., gender, age, smoking history, work habits, physical activity, skin condition, alcohol use, and medication use). Furthermore, information about disease- and treatment-related risk factors will be collected through medical records (e.g., tumor type and stage, tumor site, treatment type, etc).
General patient-, disease-, and treatment-related information | 2 weeks post-PBMT
  General and medical information will be collected through a short patient questionnaire in order to assess intrinsic risk factors (i.e., gender, age, smoking history, work habits, physical activity, skin condition, alcohol use, and medication use). Furthermore, information about disease- and treatment-related risk factors will be collected through medical records (e.g., tumor type and stage, tumor site, treatment type, etc).
Appearance and date of local and regional recurrence | 1 year follow-up post-PBMT
  The possible appearance and date of local and/or regional recurrence will be collected.
Appearance and date of local and regional recurrence | 2 year follow-up post-PBMT
  The possible appearance and date of local and/or regional recurrence will be collected.
Appearance and date of local and regional recurrence | 3 year follow-up post-PBMT
  The possible appearance and date of local and/or regional recurrence will be collected.
Appearance and date of local and regional recurrence | 4 year follow-up post-PBMT
  The possible appearance and date of local and/or regional recurrence will be collected.
Appearance and date of local and regional recurrence | 5 year follow-up post-PBMT
  The possible appearance and date of local and/or regional recurrence will be collected.
Appearance and date of secondary tumors | 1 year follow-up post-PBMT
  The possible appearance and date of secondary tumors will be collected.
Appearance and date of secondary tumors | 2 year follow-up post-PBMT
  The possible appearance and date of secondary tumors will be collected.
Appearance and date of secondary tumors | 3 year follow-up post-PBMT
  The possible appearance and date of secondary tumors will be collected.
Appearance and date of secondary tumors | 4 year follow-up post-PBMT
  The possible appearance and date of secondary tumors will be collected.
Appearance and date of secondary tumors | 5 year follow-up post-PBMT
  The possible appearance and date of secondary tumors will be collected.
Appearance and date of distant metastasis | 1 year follow-up post-PBMT
  The possible appearance and date of distant metastasis will be collected.
Appearance and date of distant metastasis | 2 year follow-up post-PBMT
  The possible appearance and date of distant metastasis will be collected.
Appearance and date of distant metastasis | 3 year follow-up post-PBMT
  The possible appearance and date of distant metastasis will be collected.
Appearance and date of distant metastasis | 4 year follow-up post-PBMT
  The possible appearance and date of distant metastasis will be collected.
Appearance and date of distant metastasis | 5 year follow-up post-PBMT
  The possible appearance and date of distant metastasis will be collected.
Date of death of any cause | 1 year follow-up post-PBMT
  If the patient dies within the first year after the treatment, their date of death will be collected.
Date of death of any cause | 2 year follow-up post-PBMT
  If the patient dies within 2 years after the treatment, their date of death will be collected.
Date of death of any cause | 3 year follow-up post-PBMT
  If the patient dies within 3 years after the treatment, their date of death will be collected.
Date of death of any cause | 4 year follow-up post-PBMT
  If the patient dies within 4 years after the treatment, their date of death will be collected.
Date of death of any cause | 5 year follow-up post-PBMT
  If the patient dies within 5 years after the treatment, their date of death will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Mebis, MD, PhD, Principal Investigator — Head of Medical Oncology Department
Locations (2):
- Belgium (2):
  - Hasselt University, Hasselt, Limburg
  - Jessa Ziekenhuis VZW, Hasselt, Limburg

IPD SHARING:
Plan to Share IPD: No